CLINICAL TRIAL: NCT02266030
Title: Effect of Cilostazol on Coronary Artery Stenosis and Plaque Characteristics in Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of Cilostazol on Coronary Artery Stenosis and Plaque Characteristics in Patients With T2DM
Acronym: ESCAPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1010/114-005
Record Dates: First submitted 2014-10-11; First posted 2014-10-16 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Cilostazol; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cilostazol (Experimental): Cilostazol 100-200 mg qd
  Interventions: Drug: Cilostazol
- Aspirin (Active Comparator): Asprin 100mg qd for active comparator
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Cilostazol — Pletaal as an active drug
  Other Names: Pletaal
  Arms: Cilostazol
Drug: Aspirin — Aspirin as an active comparator
  Arms: Aspirin

SUMMARY:
This is a prospective interventional study to assess the effect of cilostazol compared with aspirin in Korean T2DM patients with atherosclerosis.

DETAILED DESCRIPTION:
Type 2 diabetes has been increased exponentially, arousing serious economic, social and health repercussions. Also, macrovascular complications of diabetes such as myocardial infarct or stroke have been increased. Individuals with diabetes have a greater risk of cardiovascular disease (CVD), approximately two to four times than that of those without diabetes. Currently, the U.S. Food and Drug Administration requires demonstration that new anti-hyperglycemic agents do not increase CV risk. The comprehensive and multifactorial management in type 2 diabetes, which includes control of hypertension, dyslipidemia and obesity, is known to significantly reduce the risk of CVD as shown in Steno-2 study. However, most anti-diabetic agents currently used in clinical practice do not seem to provide enough CV protection.

This is a prospective interventional study to assess the effect of cilostazol compared with aspirin in Korean T2DM patients with atherosclerosis. T2DM patients who have coronary artery stenosis by MDCT at least 3 months prior to this investigation will be enrolled.

Considering drop out due to adverse events or follow up loss, sufficient patients will be enrolled. Their medical record will be reviewed and relevant clinical and laboratory findings will be collected.

Cardiac computed tomography (CT) was introduced in the early 1990s. However, electron-beam CT (EBCT) only provided information on simple coronary artery calcium score (CAC). Recently, MDCT has been introduced, which can evaluate coronary arteries comprehensively. MDCT images can provide measurements of CAC, the degree of stenosis, and the characteristics of plaque including its potential vulnerability. These findings of MDCT have been reported to be in good agreement with intravascular ultrasound.

All scans are analyzed independently by two experienced investigators using a 3D workstation, who are blinded to the clinical information (Brilliance; Philips Medical Systems). After independent evaluations are made, a consensus interpretation is arrived at regarding the final MDCT diagnosis. Each lesion is identified using a multiplanar reconstruction technique and maximum intensity projection of the short axis, in two-chamber and four-chamber views. Image quality is evaluated on a per-segment basis and classified. Plaque characteristics on a per-segment basis are analyzed according to the modified American Heart Association classification.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with HbA1c ≥ 6.0% at screening visit
* Male or female between 30 and 80 years of age
* Coronary artery stenosis: 25-75% without no evidence of acute coronary syndrome
* No history of previous myocardial infarction
* Estimated GFR ≥ 60 ml/min/1.73m²

Exclusion Criteria:

* SBP/DBP> 160/110
* Congestive heart failure
* Allegy to radiocontrast dye
* Allegy to aspirin or cilostazol
* Acute bleeding
* History of ulcer bleeding
* GOT/GPT > 100/100
* Other antiplatlet medication

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Coronary artery stenosis | one year
  Severity of coronary artery stenosis (%)

SECONDARY OUTCOMES:
Plaque characteristics | one year
  Noncalified plaque
Plaque characteristics | one year
  Mixed plaque
Plaque characteristics | one year
  Calcified plaque
Multivessel involvement | one year
  Multivessel involvement in coronary arteries
Main vessel involvement | one year
  Left main and/or proximal LAD stenosis
Coronary artery calcium (CAC) score | one year
  Agatston score for CAC
Glucose homeostasis | one year
  Changes in HbA1c
Glucose homeostasis | one year
  Changes in fasting glucose concentration
Lipid metabolism | one year
  Changes in TG concentration
Lipid metabolism | one year
  Changes in HDL-concentration concentration

OTHER OUTCOMES:
Bleeding risk | one year
  Any type of bleeding
Headache | one year
  Any type of headache
Heart rate | one year
  Frequence of heart beat per min

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD, PhD, Principal Investigator — SNUBH
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Bundang-gu, South Korea